CLINICAL TRIAL: NCT05230238
Title: Pituitary Gland Stimulation for Cancer Pain Relief
Acronym: PGS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, wrvanfurth, neurosurgeon, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P21.036
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Oncology Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pituitary stimulation (Experimental): Patients will receive pituitary stimulation as oncology pain treatment.
  Interventions: Device: Pituitary gland stimulation

INTERVENTIONS:
Device: Pituitary gland stimulation — Pituitary gland stimulation via an surface electrode connected to an external neurostimulator

SUMMARY:
Patients will undergo an implantation of an extradural pituitary surface electrode in the pituitary fossa. The electrode will be attached to a neurostimulator via which the patient will receive up to 8 (patient requested) stimulations per day.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* In palliative phase of metastatic disease, without options for further systemic treatment or radiotherapy
* Inadequately controlled pain with standard care
* Most prominent part of experienced pain is nociceptive
* Karnofsky Performance Score ≥30

Exclusion Criteria:

* Not fit for general anesthesia
* Pregnancy
* Unfavorable local anatomy for PGS, due to a disease process, or anatomical configuration
* Clinical signs of posterior pituitary gland disfunction
* Recent history of alcohol or drug abuse
* Severe immunodeficiency
* Need for anticoagulation therapy that cannot be abrogated for surgery
* Need for subsequent MRI-imaging
* Cognitive impairments prohibiting full understanding of study and ability to provide informed consent
* Not able to adequately communicate in Dutch or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Perceived pain | 4 months
  Numeric Rating Scale (0= no pain, 10=most severe pain)
Pain Medication | 4 months
  Morphine Equivalent Doses for background and escape medication

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Furth, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided